CLINICAL TRIAL: NCT04335123
Title: An Open Label Phase 1 Trial of Losartan for Worsening Respiratory Illness in COVID-19
Brief Title: Study of Open Label Losartan in COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Matthias Salathe, MD, Professor- University of Kansas Medical Center, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00145514
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; losartan; respiratory failure; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: 30 patients with COVID-19 and respiratory failure who meet criteria and agree to participation in the study will be placed on losartan 25 mg once daily on study day 0. If parameters are met the dose of losartan will be increased to 50 mg once daily on study day 3. Patients and/or surrogate decision maker who do not give consent to treatment will be asked to allow collection of data from their medical record for use as a control group. We will also collect medical information relating to safety criteria on historical controls treated at the University of Kansas Hospital in the 30 days prior to the study start date and during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Label Losartan (Experimental): 50 patients with COVID-19 and respiratory failure who meet criteria and agree to participation in the study will be placed on losartan 25 mg once daily on study day 0. If parameters are met the dose of losartan will be increased to 50 mg once daily on study day 3. Participants will continue losartan until they experience resolution of respiratory failure (normal oxygen levels on room air), are discharged from the hospital, meet stoppage criteria or complete 14 days of therapy.
  Interventions: Drug: Losartan
- External Control (No Intervention): Matched - contemporaneous control who met enrollment criteria and were treated at UKHS during the COVID-19 pandemic period.

INTERVENTIONS:
Drug: Losartan — 25 mg QD from day 0 to day 3. Dose escalation to 50 mg QD until study completion
  Other Names: Cozaar
  Arms: Open Label Losartan

SUMMARY:
This is an open label, phase 1 clinical trial to evaluate the safety of losartan in respiratory failure due to COVID-19.

Briefly, 34 patients with COVID-19 and respiratory failure who meet eligibility criteria and agree to participation in the study will be placed on losartan 25 mg daily on study day 0. If parameters are met the dose of losartan will be increased to 50 mg once daily on study day 3. Participants will continue losartan until they experience resolution of respiratory failure (normal oxygen levels on room air), are discharged from the hospital, meet stoppage criteria (detailed below) or complete 14 days of therapy.

Patients and/or surrogate decision maker who do not give consent to treatment will be asked to allow collection of data from their medical record for use as a control group. We will also collect medical information relating to safety criteria on historical controls treated at the University of Kansas Hospital in the 30 days prior to the study start date and during the study period.

DETAILED DESCRIPTION:
This is an open label, phase 1 clinical trial to evaluate the safety of losartan in respiratory failure due to COVID-19.

Clinical Trial setup:

Detailed inclusion and exclusion criteria are listed below. Briefly, 34 patients with COVID-19 and respiratory failure who meet criteria and agree to participation in the study will be placed on losartan 25 mg daily on study day 0. If parameters are met the dose of losartan will be increased to 50 mg once daily on study day 3. Participants will continue losartan until they experience resolution of respiratory failure (normal oxygen levels on room air), are discharged from the hospital, meet stoppage criteria (detailed below) or complete 14 days of therapy.

Patients and/or surrogate decision maker who do not give consent to treatment will be asked to allow collection of data from their medical record for use as a control group.

Stoppage criteria for losartan

* Hyperkalemia (persistent values >5.5 mM recorded on at least 2 readings).
* Worsening renal function (Cockcroft-Gault <30 mL/min/1.73 m2) or urinary output <20 mL/h.
* Skin rashes, palpitations or other moderate or severe adverse events (interference with usual daily activities) without clear explanation should warrant immediate cessation of treatment and notification of study personnel.
* Development of sustained hypotension defined as SBP <90 mmHg, DBP <60 mmHg recorded on at least two readings 30 min apart or use of norepinephrine >0.1 µg/kg/min.
* Any change in monitor lab parameters deemed significant and potentially related to study drug by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years admitted to the University of Kansas Health System.
* Confirmation of infection with SARS-CoV-2 by PCR testing.
* Hypoxic respiratory failure Requiring mechanical ventilation or oxygen OR a SpO2 ≤94% on room air or a PaO2/FiO2 (P/F) ratio <300 OR tachypnea (respiratory rate ≥24 breaths/min). Criteria to be met within 48 hours prior to Day 0.
* Other concomitant medications such as antivirals and hydroxychloroquine are allowed.
* Participants prescribed standard of care (SOC) losartan (25mg QD) within 48 hours of consenting may be considered for enrollment if eligibility criteria are met based on EMR data assessment, i.e. no other ARB or ACE prior to SOC medication administration. If participant is eligible and signs consent form, investigational losartan 25mg QD will be ordered to replace SOC prescription on the following scheduled dose.

Exclusion Criteria:

* Pregnancy.
* Respiratory failure due to a process other than COVID-19.
* Intolerance to ARBs.
* Previous treatment with an ARB or ACE inhibitor (see exception in inclusion criteria).
* Current chronic use of medication with known interactions with losartan including NSAIDs (intermittent prior use is acceptable), potassium supplementation aliskiren.
* Blood pressure less than 90 mm Hg systolic or 60 mm Hg diastolic recorded on at least two readings 30 min apart.
* Need for vasopressors, unless norepinephrine ≤0.1 µg/kg/min
* Hyperkalemia (serum K+ >5.5 mM).
* Known cardiac failure (left ventricular ejection fraction ≤35%), renal insufficiency (Cockcroft-Gault <30 mL/min/1.73 m2 or urinary output <20 mL/h), hepatic failure (LFTs > 5x normal upper limit).
* Known renal artery stenosis.
* Neurological, psychiatric, endocrine or neoplastic diseases that are judged to interfere with participation in the study.
* On another interventional trial (including one for COVID-19) that excludes participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Salathe, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposals should be directed to msalathe@kumc.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Smolander J, Bruchfeld A. [COVID-19 and kidney disease]. Lakartidningen. 2020 Jul 13;117:20110. Swedish. PMID 32658300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: External control group were hospitalized during study period and met enrollment criteria and were not enrolled. Participants were matched to losartan group on baseline characteristics.
Groups:
- Open Label Losartan: 34 patients with COVID-19 and respiratory failure participated in the study and were placed on losartan 25 mg once daily on study day 0. Losartan dose was increased to 50 mg once daily on study day 3. Participants continued losartan until they experienced resolution of respiratory failure (normal oxygen levels on room air), were discharged from the hospital, met stoppage criteria or completed 14 days of therapy.
  Losartan: 25 mg QD from day 0 to day 3. Dose escalation to 50 mg QD until study completion
- External Control: A group of external controls matched to the enrolled participants
Period: Overall Study
Arm/Group | Open Label Losartan | External Control
Started | 34 | 46
Completed | 30 | 46
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- External Controls: 46 external controls matched to losartan participants upon baseline characteristics.
- Total: Total of all reporting groups
Arm/Group | Open Label Losartan | External Controls | Total
Number analyzed (Participants) | 30 | 46 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (15.1) | 53.8 (15.5) | 54 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 34
  Male | 17 | 25 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 21 | 29
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by Protocol Definition of AE
Description: Safety will be reported based on Protocol defined AEs.
  For the purpose of this protocol, an AE will be defined as as any untoward medical occurrence in a subject during the study listed under DMSB - Anticipated Adverse Events and Grading Scale section of this protocol as well as safety monitoring data listed on protocol table 1 as well as stoppage criteria for losartan.
  The event does not necessarily have a causal relationship with the treatment. AEs will be collected for both study groups, treatment and control from the time the ICF is signed until the subject completes study participation.
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 24 | 44

2. Secondary Outcome: Number of Days on Supplemental Oxygen in Respiratory Failure Due to COVID-19
Description: Number of days on supplemental oxygen in respiratory failure due to COVID-19
Time Frame: 14 days of losartan treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
days | 4 [2 to 6] | 4 [0 to 9]

3. Secondary Outcome: Number of Participants With Mechanical Ventilation Use
Description: Number of participants with mechanical ventilation use
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 2 | 9

4. Secondary Outcome: Days on Mechanical Ventilation
Description: Days on mechanical ventilation
Time Frame: 14 days of losartan treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
days | 0 [0 to 0] | 11 [8 to 14]

5. Secondary Outcome: Number of Participants With Non-invasive Positive Pressure Ventilation or Heated High Flow Nasal Cannula Use
Description: Number of participants with non-invasive positive pressure ventilation or heated high flow nasal cannula use
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 6 | 3

6. Secondary Outcome: Days on Non-invasive Positive Pressure Ventilation or High Flow Nasal Cannula
Description: Days on non-invasive positive pressure ventilation or high flow nasal cannula
Time Frame: 14 days of losartan treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
days | 0 [0 to 0] | 5 [3.5 to 7.5]

7. Secondary Outcome: Number of Participants With Transfer to ICU From Non-ICU Hospital Bed
Description: Number of participants with transfer to ICU from non-ICU hospital bed
Time Frame: 14 days of losartan treatment
Population: Data regarding transfer to ICU was not collected for any participants during study period and thus not reported.
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: ICU Length of Stay (Days)
Description: ICU length of stay (days)
Time Frame: 14 days of losartan treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
days | 0 [0 to 11.5] | 10 [7.5 to 13.5]

9. Secondary Outcome: in Hospital Mortality Rate
Description: in hospital mortality rate
Time Frame: 14 days after study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 1 | 3

10. Secondary Outcome: Hospital Length of Stay (Days)
Description: Hospital length of stay (days)
Time Frame: from enrollment through hospital discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
days | 9 [6 to 14.75] | 7 [4 to 13.5]

11. Secondary Outcome: Cumulative Number of Participants With of Severe Adverse Events
Description: Cumulative number of participants with severe adverse events
Time Frame: 14 days of losartan treatment
Measure: Number; unit: participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
participants | 0 | 0

12. Secondary Outcome: Number of Participants With Increase of Supplemental Oxygen Needs From Baseline.
Description: Number of participants with increase in supplemental oxygen needs from baseline.
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 4 | 12

13. Secondary Outcome: Number of Participants With Medications With Possible Antiviral Activity (Hydroxychloroquine, Lopinavir/Ritonavir, Ribavirin or Remdesivir) or Adjunctive Therapy Use (e.g., Tocilizumab)
Description: Number of participants with medications with possible antiviral activity (hydroxychloroquine, lopinavir/ritonavir, ribavirin or remdesivir) or adjunctive therapy use (e.g., tocilizumab)
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 30 | 30

14. Secondary Outcome: Number of Participants With Extracorporeal Membrane Oxygenation Use
Description: Number of participants with extracorporeal membrane oxygenation use
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Renal Replacement Therapy Use
Description: Number of participants with renal replacement therapy use
Time Frame: 14 days of losartan treatment
Population: This outcome was not collected for study participants, thus results are not reported
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With Intolerance to High Dose (50mg) Losartan After Tolerating 25mg
Description: Number of participants with intolerance to high dose (50mg) losartan after tolerating 25mg
Time Frame: 14 days of losartan treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Losartan | External Controls
Number analyzed (Participants) | 30 | 46
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: From enrollment to hospital discharge, up to day 14.
Arm/Group | Open Label Losartan | External Controls
All-Cause Mortality (participants affected / at risk) | 1/30 | 3/46
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/46
Other Adverse Events (participants affected / at risk) | 24/30 | 44/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Losartan (N=30) | External Controls (N=46)
Low hemoglobin (Blood and lymphatic system disorders) | 15 (15) | 32 (32)
Elevated AST (Hepatobiliary disorders) | 11 (11) | 30 (30)
Elevated ALT (Hepatobiliary disorders) | 12 (12) | 23 (23)
Elevated creatinine (Renal and urinary disorders) | 9 (9) | 12 (12)
hypotension (Vascular disorders) | 8 (8) | 14 (14)
Elevated Alkaline phosphatase (Hepatobiliary disorders) | 5 (5) | 14 (14)
Elevated potassium (Renal and urinary disorders) | 3 (3) | 14 (14)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 14 (14)
Low platelets (Blood and lymphatic system disorders) | 1 (1) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04335123/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04335123/ICF_001.pdf